CLINICAL TRIAL: NCT06223477
Title: Evaluation of the Effects of Platelet-rich Fibrin and Vitamin Dꝫ Injections on the Periodontal Health During Canine Distalization: A Randomized Controlled Clinical Trial
Brief Title: Effects of Platelet-rich Fibrin and Vitamin Dꝫ Injections on the Periodontal Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Rehab Abd El Razek Abd El Aziz Khalil, Lecturer of Orthodontics, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: # REC-FDBSU/P106042023-03/AR
Record Dates: First submitted 2023-12-27; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Health
Keywords: platelet-rich fibrin; vitamin D3; periodontal health
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: split-mouth, prospective, single-center, single-blinded, two-arm randomized clinical trial with a 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: Single-blinded limited to the outcome assessment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-rich Fibrin (Experimental): A 20 ml blood sample will be drawn from the median cubital vein into a PRF tube. Centrifugation will be done at 700 rpm for 3 minutes and the liquid of PRF will be suctioned out using a separate syringe. PRF will be injected distal to the canine on the experimental side three times; at the beginning of canine retraction (T0), 1 month after the start of canine retraction (T1), and 2 months after the start of canine retraction (T2).
  Interventions: Other: Platelet-rich Fibrin
- Vitamin D3 (Experimental): Subjects will receive vitamin Dꝫ injection distal to the canine on the experimental side three times; at the beginning of canine retraction (T0), 1 month after the start of canine retraction (T1), and 2 months after the start of canine retraction (T2).
  Interventions: Other: Vitamin D3

INTERVENTIONS:
Other: Platelet-rich Fibrin — PRF will be injected distal to the canine on the experimental side.
  Arms: Platelet-rich Fibrin
Other: Vitamin D3 — Vitamin Dꝫ will be injected distal to the canine on the experimental side
  Arms: Vitamin D3

SUMMARY:
The study aims to evaluate the effect of using PRF and vitamin Dꝫ injections on periodontal health and parameters and compare them when used to facilitate orthodontic treatment.

DETAILED DESCRIPTION:
* Participants will be recruited from the Faculty of Dentistry, Beni-Suef University. All subjects will be informed of the treatment procedures and will sign a consent form.
* Subjects will be randomly divided into two groups:

Group 1 (PRF group): upper canine retraction will be facilitated by PRF injection that will be randomly assigned to one side (experimental side). The contralateral side will serve as the control one.

Group II (Vitamin Dꝫ group): canine retraction will be facilitated by Vitamin Dꝫ injection that will be randomly assigned to one side (experimental side). The contralateral side will serve as the control one.

* The predicted sample size (n) was a total of (28) cases (i.e. 14 cases per group). Sample size calculation was performed using G*Power version 3.1.9.7
* Simple randomization will be designed with the aid of a computer-generated schedule with 1:1 allocation ratio. Allocation concealment will be achieved using identical opaque, sealed envelopes. Randomization and allocation concealment will be performed by one of the academic staff who will not be involved in the study and will keep the allocation table away from the operators. The operator will shuffle the sealed envelopes and will ask the patient to pick one envelope at the time of recruitment. In each group, a randomly selected side will act as the experimental side while the contralateral side will serve as the control. Blinding of the operators will not be applicable and so blinding will be limited to the outcome assessment.

Methodology:

* All patients will be treated with a 0.022-inch MBT bracket system. Leveling and alignment phase will be completed until a 0.017 X 0.025''stainless steel wire will be inserted passively into the bracket slot. Before canine retraction, the subject will be randomly assigned to one of the groups (PRF or Vitamin Dꝫ group). In both groups, canine retraction will be performed with closed Ni-Ti coil springs with a force of 150 g per side that will be adjusted by the use of a force gauge.

ELIGIBILITY:
Inclusion criteria:

1. Age: 18- 40 years old.
2. Angle Class I or Class II dental malocclusion that required bilateral maxillary first premolar extraction and upper canine retraction as a part of the treatment plan.
3. Good to fair oral hygiene.
4. Normal probing depth.

Exclusion criteria:

1. Active periodontal disease.
2. Poor oral hygiene.
3. Systemic diseases or medications that alter bone metabolism or tooth movement.
4. Craniofacial anomalies.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of using PRF and Vitamin Dꝫ injections on periodontal health and compare them. | 3 - 4 months
  Clinical periodontal examination of the upper canines will be done before and after retraction on the experimental and control sides by recording the probing depth (PD).
  • The probing depth will be measured from the gingival margin to the base of the gingival sulcus in millimeters by using a manual periodontal probe (William's probe). The measurements will be recorded at 6 sites around the tooth.

SECONDARY OUTCOMES:
Investigate the effect of PRF and Vitamin Dꝫ injections on the gingival thickness. | 3 - 4 months
  The gingival thickness will be recorded using an endodontic file with a stopper, which is placed horizontally, perpendicular to the long axis of the tooth on the labial gingiva.

OTHER OUTCOMES:
Evaluate the effect of using PRF and Vitamin Dꝫ injections on the width of keratinized mucosa (KM) | 3 - 4 months
  The width of keratinized mucosa (KM) on the facial aspect will be measured in millimeters at the mid-facial aspects from the mucogingival junction to the free gingival margin using a periodontal probe before and after canine retraction.
Evaluate the effect of using PRF and Vitamin Dꝫ injections on the gingival index. | 3 - 4 months
  The gingival index will be evaluated by the following scores before and after canine retraction:
  0: Normal gingival, no inflammation, no discoloration, no bleeding.
  1. Mild inflammation, slight color change, mild alteration of gingival surface, no bleeding.
  2. Moderate inflammation, erythema, swelling, bleeding on probing or when pressure is applied
  3. severe inflammation, severe erythema, swelling, tendency towards spontaneous bleeding some ulceration.
Evaluate the effect of using PRF and Vitamin Dꝫ injections on the plaque index. | 3 - 4 months
  Plaque index will be evaluated by the following scores before and after canine retraction:
  0: No dental plaque
  1. Thin film of plaque at the gingival margin not visible by naked eye and detect by probe
  2. Moderate film of plaque at the gingival margin, interdental space free of plaque visible by naked eye
  3. Heavy plaque accumulation at the gingival margin on interdental space filled with plaque (calculus)
Evaluate the effect of using PRF and Vitamin Dꝫ injections on the clinical attachment level (CAL) | 3 - 4 months
  Clinical attachment level (CAL) will be measured from the cementoenamel junction to the base of the periodontal pocket in millimeters by using a periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Khalil, Principal Investigator — Faculty of Dentistry Beni Suef University
Locations (1):
- Faculty of Dentistry Beni Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta P, Bhagyalakshmi A, Avinash BS, Prashant A, Raghunath N. Evaluation of injectable platelet-rich fibrin effect on the rate of canine retraction and alkaline phosphatase levels: An in-vivo study. Am J Orthod Dentofacial Orthop. 2022 Nov;162(5):735-743. doi: 10.1016/j.ajodo.2021.07.019. Epub 2022 Aug 23. PMID 36008239
- [Background] Cagli Karci I, Baka ZM. Assessment of the effects of local platelet-rich fibrin injection and piezocision on orthodontic tooth movement during canine distalization. Am J Orthod Dentofacial Orthop. 2021 Jul;160(1):29-40. doi: 10.1016/j.ajodo.2020.03.029. Epub 2021 May 4. PMID 33962809
- [Background] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Effect of injectable platelet-rich fibrin (i-PRF) in accelerating orthodontic tooth movement : A randomized split-mouth-controlled trial. J Orofac Orthop. 2021 Jul;82(4):268-277. doi: 10.1007/s00056-020-00275-x. Epub 2021 Jan 22. PMID 33481053
- [Background] Varughese ST, Shamanna PU, Goyal N, Thomas BS, Lakshmanan L, Pulikkottil VJ, Ahmed MG. Effect of Vitamin D on Canine Distalization and Alveolar Bone Density Using Multi-slice Spiral CT: A Randomized Controlled Trial. J Contemp Dent Pract. 2019 Dec 1;20(12):1430-1435. PMID 32381845
- [Background] Bollen AM, Cunha-Cruz J, Bakko DW, Huang GJ, Hujoel PP. The effects of orthodontic therapy on periodontal health: a systematic review of controlled evidence. J Am Dent Assoc. 2008 Apr;139(4):413-22. doi: 10.14219/jada.archive.2008.0184. PMID 18385025
- [Background] Faour NH, Dayoub S, Hajeer MY. Evaluation of the Hyaluronic Acid Versus the Injectable Platelet-Rich Fibrin in the Management of the Thin Gingival Phenotype: A Split-Mouth Randomized Controlled Clinical Trial. Cureus. 2022 May 18;14(5):e25104. doi: 10.7759/cureus.25104. eCollection 2022 May. PMID 35607316
- [Background] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Three-dimensional evaluation of the effects of injectable platelet rich fibrin (i-PRF) on alveolar bone and root length during orthodontic treatment: a randomized split mouth trial. BMC Oral Health. 2021 Mar 2;21(1):92. doi: 10.1186/s12903-021-01456-9. PMID 33653326
- [Background] Lu EM. The role of vitamin D in periodontal health and disease. J Periodontal Res. 2023 Apr;58(2):213-224. doi: 10.1111/jre.13083. Epub 2022 Dec 20. PMID 36537578